CLINICAL TRIAL: NCT01218542
Title: Whole Brain Radiation Therapy With Simultaneous Boost to Gross Metastatic Tumor Volume Using Volumetric Modulated Arc Therapy (RapidArc)
Brief Title: Whole Brain Radiation Therapy With Boost to Metastatic Tumor Volume Using RapidArc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Hui-Kuo Shu, MD, PhD, MD, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00045035; WCI1784-10 (Other: Other)
Record Dates: First submitted 2010-09-30; First posted 2010-10-11 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Neoplasm Metastasis
Keywords: Secondary brain malignancies; RapidArc; Volumetric modulated arc therapy
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Volumetric modulated arc therapy (Experimental): Single arm pilot study treating patients with 25 Gy in 10 fractions to the whole brain with simultaneous infield boost (SIB) to a total of 45 Gy in 10 fractions to gross brain metastatic disease.
  Interventions: Radiation: Volumetric modulated arc therapy

INTERVENTIONS:
Radiation: Volumetric modulated arc therapy — Using volumetric modulated arc therapy to give simultaneous infield boost to gross metastatic brain lesions during whole brain radiation therapy.

SUMMARY:
Brain metastases are the most common adult intracranial tumor, occurring in approximately 10% to 30% of adult cancer patients, and represent an important cause of morbidity and mortality. The most widely used treatment for patients with multiple brain metastases is whole brain radiation therapy (WBRT). The use of WBRT after resection or stereotactic radiosurgery (SRS) has been proven to be effective in terms of improving local control of brain metastases.

RapidArc (RA) (Varian Medical Systems, Palo Alto, CA) is a new method of delivering radiation that uses "arcs" to deliver highly conformal intensity modulated three dimensional dose distributions. The purpose of this investigation is to evaluate an alternative strategy for giving WBRT with highly focal boost to gross visible lesions in patients with brain metastasis.

Given the limitations of the SRS boost technique, the purpose of our investigation is to evaluate an alternative strategy for giving WBRT with highly focal boost to gross visible lesions in patients with brain metastasis. In this study, we plan to assess the tolerability of using volumetric modulated arc therapy (RapidArc) on patients with brain metastasis to simultaneously treat the entire brain with a concomitant focal boost to grossly identified lesions on MRI scan to try to improve local control and reduce neurocognitive toxicities.

This previous version of this study was a phase I dose escalation trial giving 25 Gy in 10 fractions to the whole brain with simultaneous infield boost (SIB) to a total of 45 Gy in 10 fractions to gross brain metastatic disease. Prior to this, patients were enrolled onto one of two cohorts with whole brain dose of 30 Gy in 10 fractions with SIB to total of 45 Gy in 10 fractions to gross brain metastatic disease or whole brain dose of 37.5 Gy in 15 fractions with SIB to total of 52.5 Gy in 15 fractions to gross brain metastatic disease. A total of 12 patients have been previously enrolled on this trial. No patients have experienced a dose limiting toxicity (grade 3 or above) at least possibly due to study therapy. Also, no patients experienced local brain failure/progression at a site of treated metastatic brain disease. Based on this, we no longer feel that dose escalation to the gross brain disease is warranted and would proceed with a single arm pilot study treating patients with 25 Gy in 10 fractions to the whole brain with simultaneous infield boost (SIB) to a total of 45 Gy in 10 fractions to gross brain metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic proven diagnosis of solid tumor malignancy.
* Age ≥ 18.
* KPS ≥ 70.
* Mini Mental Status Exam (MMSE) ≥ 18 prior to study entry.
* RPA class I (KPS ≥ 70, primary cancer controlled, age < 65, metastases in brain only) or class II (lack of one or more of class I criteria).
* One to ten brain metastatic lesions.

Exclusion Criteria:

* Previous whole brain radiation therapy.
* Previous radiosurgery to any currently progressive gross metastatic disease.
* Previous radiosurgery to any intracranial site within the prior 6 weeks.
* Recursive partitioning analysis (RPA) class III (KPS < 70).
* Radiosensitive (eg. small cell lung carcinomas, germ cell tumors, leukemias, or lymphomas) or unknown tumor histologies.
* Concurrent chemotherapy (no chemotherapy starting 14 days before start of radiation).
* Evidence of leptomeningeal disease by MRI and/or cerebrospinal fluid (CSF) cytology.
* Current pregnancy.
* No metastases to brain stem, midbrain, pons, or medulla or within 7 mm of the optic apparatus (optic nerves and chiasm).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-09-22 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Kuo Shu, MD, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zimm S, Wampler GL, Stablein D, Hazra T, Young HF. Intracerebral metastases in solid-tumor patients: natural history and results of treatment. Cancer. 1981 Jul 15;48(2):384-94. doi: 10.1002/1097-0142(19810715)48:23.0.co;2-8. PMID 7237407
- [Background] Sundstrom JT, Minn H, Lertola KK, Nordman E. Prognosis of patients treated for intracranial metastases with whole-brain irradiation. Ann Med. 1998 Jun;30(3):296-9. doi: 10.3109/07853899809005858. PMID 9677016
- [Background] CHAO JH, PHILLIPS R, NICKSON JJ. Roentgen-ray therapy of cerebral metastases. Cancer. 1954 Jul;7(4):682-9. doi: 10.1002/1097-0142(195407)7:43.0.co;2-s. No abstract available. PMID 13172684
- [Background] Gaspar L, Scott C, Rotman M, Asbell S, Phillips T, Wasserman T, McKenna WG, Byhardt R. Recursive partitioning analysis (RPA) of prognostic factors in three Radiation Therapy Oncology Group (RTOG) brain metastases trials. Int J Radiat Oncol Biol Phys. 1997 Mar 1;37(4):745-51. doi: 10.1016/s0360-3016(96)00619-0. PMID 9128946
- [Background] Patchell RA, Regine WF. The rationale for adjuvant whole brain radiation therapy with radiosurgery in the treatment of single brain metastases. Technol Cancer Res Treat. 2003 Apr;2(2):111-5. doi: 10.1177/153303460300200206. PMID 12680791
- [Background] Arbit E, Wronski M, Burt M, Galicich JH. The treatment of patients with recurrent brain metastases. A retrospective analysis of 109 patients with nonsmall cell lung cancer. Cancer. 1995 Sep 1;76(5):765-73. doi: 10.1002/1097-0142(19950901)76:53.0.co;2-e. PMID 8625178
- [Background] Andrews DW, Scott CB, Sperduto PW, Flanders AE, Gaspar LE, Schell MC, Werner-Wasik M, Demas W, Ryu J, Bahary JP, Souhami L, Rotman M, Mehta MP, Curran WJ Jr. Whole brain radiation therapy with or without stereotactic radiosurgery boost for patients with one to three brain metastases: phase III results of the RTOG 9508 randomised trial. Lancet. 2004 May 22;363(9422):1665-72. doi: 10.1016/S0140-6736(04)16250-8. PMID 15158627
- [Background] Lagerwaard FJ, van der Hoorn EA, Verbakel WF, Haasbeek CJ, Slotman BJ, Senan S. Whole-brain radiotherapy with simultaneous integrated boost to multiple brain metastases using volumetric modulated arc therapy. Int J Radiat Oncol Biol Phys. 2009 Sep 1;75(1):253-9. doi: 10.1016/j.ijrobp.2009.03.029. Epub 2009 Jul 4. PMID 19577856
- [Background] Bauman G, Yartsev S, Fisher B, Kron T, Laperriere N, Heydarian M, VanDyk J. Simultaneous infield boost with helical tomotherapy for patients with 1 to 3 brain metastases. Am J Clin Oncol. 2007 Feb;30(1):38-44. doi: 10.1097/01.coc.0000245473.41035.c4. PMID 17278893
- [Result] Zhong J, Waldman AD, Kandula S, Eaton BR, Prabhu RS, Huff SB, Shu HG. Outcomes of whole-brain radiation with simultaneous in-field boost (SIB) for the treatment of brain metastases. J Neurooncol. 2020 Mar;147(1):117-123. doi: 10.1007/s11060-020-03405-y. Epub 2020 Jan 22. PMID 31970594

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at Winship Cancer Institute of Emory University from September 2010 to September 2015.
Period: Overall Study
Arm/Group | Volumetric Modulated Arc Therapy
Started | 22
Completed | 13
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Volumetric Modulated Arc Therapy
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Locoregional Control of Treating Brain Metastasis Patients
Description: The cumulative incidences of recurrence locally and in the whole brain were reported at the patient level.
Time Frame: Locoregional control at 1 year
Population: Feasibility by our criteria was met for all participants.
Measure: Number; unit: percentage of participants
Arm/Group | Volumetric Modulated Arc Therapy
Number analyzed (Participants) | 13
percentage of participants
  1-year Local Control | 92
  Lesion Level Control | 98.6
  1-year Regional Control | 46
  Intracranial Control | 46
  Distant Intracranial Recurrence | 87.5

2. Secondary Outcome: Brain Progression-free Survival
Description: Defined as period of time from study entry to to death from any cause or brain tumor recurrence or progression.
Time Frame: 11 months median follow up period.
Measure: Median (Full Range); unit: months
Arm/Group | Volumetric Modulated Arc Therapy
Number analyzed (Participants) | 13
months | 5.7 [2.9 to 26.2]

3. Secondary Outcome: Overall Survival
Description: Defined time from study entry to death from any cause.
Time Frame: 11 months median follow up period.
Measure: Median (Full Range); unit: months
Groups:
- Volumetric Modulated Arc Therapy: The 2-year neurocognitive effect was not collected. We collected and reported neurocognitive data up to 6 months after treatment.
Arm/Group | Volumetric Modulated Arc Therapy
Number analyzed (Participants) | 13
months | 8.6 [4.1 to 29.6]

4. Secondary Outcome: Neurocognitive Effects
Description: Neurological test score were assessed using the Hopkins Verbal Learning Test-Revised (HVLT).
  In the HVLT 12 words are read and the participant is asked to recall them, this is completed 3 times.
  Total words recalled are summed to give a score for Total Recall (0-36, higher scores demonstrated better recall).
  Delayed recall is conducted 20-25 minutes later on the same list of 12 words (scored 0-12 with higher scores demonstrating better recall).
  Retention is calculated as the percent of words recalled (scored 0-100, higher scores representing better recall).
  Recognition Discrimination is tested by a series of yes/no responses from the participant identifying 12 target words from a list of 24 and calculated by the number of true positives minus the number of true negatives with higher scores indicating a better outcome.
Time Frame: 11 months median follow up period.
Measure: Mean (95% Confidence Interval); unit: fraction of post-tx over pre-tx scores
Arm/Group | Volumetric Modulated Arc Therapy
Number analyzed (Participants) | 13
fraction of post-tx over pre-tx scores
  Total Recall | 1.0 [0.73 to 1.27]
  Delayed Recall | 1.09 [0.90 to 1.28]
  Retention | 0.99 [0.72 to 1.258]
  Recognition Discrimination | 0.96 [0.77 to 1.14]

5. Secondary Outcome: Quality of Life as Measured by the FACT-Br Subscales
Description: The Functional Assessment of Cancer Therapy-Brain (FACT-Br) were summed to create the FACT brain trial outcome index (FACT-BR TOI), FACT general (FACT-G), and FACT brain total (FACT-BR Total).
  Three FACT scales were calculated. The higher the value the better the score, i.e., the better the quality of life perceived by patient.
  FACT BR TOTAL (FACT-G + BrCS, possible range 0 - 200) FACT-BR TOI (Trial Outcome Index = Physical Well Being _ Functional Well Being +BrCS, possible range 0 - 148) FACT-G (Fact General, possible range 0 - 108)
Time Frame: 11 month median follow up
Measure: Mean (95% Confidence Interval); unit: fraction of post-tx over pre-tx scores
Arm/Group | Volumetric Modulated Arc Therapy
Number analyzed (Participants) | 13
fraction of post-tx over pre-tx scores
  FACT-BR Total | 1.0 [0.93 to 1.08]
  FACT-BR TOI | 0.98 [0.87 to 1.081]
  FACT-G | 0.98 [0.73 to 1.23]

ADVERSE EVENTS:
Time Frame: Adverse events were collected thorughout the study assessed up to 2 year follow-up
Arm/Group | Volumetric Modulated Arc Therapy
All-Cause Mortality (participants affected / at risk) | 10/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Volumetric Modulated Arc Therapy (N=13)
Radiation Necrosis (General disorders) | 2 (2)
Fatigue (General disorders) | 8 (8)
Nausea (General disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-09): https://cdn.clinicaltrials.gov/large-docs/42/NCT01218542/Prot_SAP_000.pdf